CLINICAL TRIAL: NCT00501189
Title: Gardasil Vaccination as Therapy in Low Grade Cervical Abnormalities
Status: Withdrawn | Type: Observational
Why Stopped: recruiting issues
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dean A. Seehusen, Physician, Eisenhower Army Medical Center
Other Study IDs: DDEAMC 07-43X
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2024-06-11 (Actual); Status verified 2008-07

CONDITIONS: Papillomavirus Infections
Keywords: Gardasil; Human Papilloma Virus; Papanicolaou Smear; ASCUS; LGSIL; Human Papilloma Virus Vaccine; Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections; Atypical Squamous Cells of the Cervix | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Those getting Gardasil vaccination for low grade Pap abnormality.
  Interventions: Biological: human papillomavirus vaccine L1, type 6,11,16,18
- 2: Historical group that did not get Gardasil.

INTERVENTIONS:
Biological: human papillomavirus vaccine L1, type 6,11,16,18 — Subjects are those getting gradasil vaccination already. This is really not an intervention
  Groups: 1

SUMMARY:
This project will compare the rate of regression of minimally abnormal Pap smears to normal in women who receive Gardasil to a historical control group.

Research hypothesis: Women with low grade cervical dysplasia on Papanicolaou (Pap) smear that receive Gardasil vaccination will revert to a normal within one year at a rate 33% higher than historical controls that did not receive Gardasil vaccination.

DETAILED DESCRIPTION:
This study is looking for additional clinical outcomes in women who are already getting the Gardasil vaccination. We are not giving the vaccination as part of the research protocol. This point will be stressed to patients. Their participation or non-participation will not impact their ability to receive the vaccine series. Their participation only impacts whether or not we will contact them in the future and whether or not we will review their medical records.

Subjects will be enrolled into the study at the time of their presentation for colposcopy in the EAMC Family Medicine Clinic. Subjects will be screened for inclusion and exclusion criteria. Those found eligible will be consented for enrollment by one of the study investigators. Colposcopy records will also be searched for patients seen in the colposcopy clinic between the availability of Gardasil and the beginning of this study. Any patients who meet enrollment criteria will be contacted by phone and invited to participate in the study. These patients will be followed in the exact same way as patients enrolled upon presenting for the first time to the colposcopy clinic.

Patients will be given their first vaccination at the time of their colposcopy appointment unless they have already begun the vaccine series. Phone and email will be used to remind patients when they are due for their second and third vaccinations. Any study subject that does not receive the their 2nd or 3rd vaccine will be considered "partially vaccinated". They will not be removed from the protocol, however, because an intention-to-treat analysis is planned.

Study subjects will be followed prospectively for up to 15 months. 15 months was chosen because some patients may be late getting their one-year follow ups. AHLTA records and colposcopy clinic convenience files will be reviewed for each patient periodically. Patients who meet criteria to return to routine annual Pap smear, based on ASCCP guidelines, during the next 11 to 15 months will be considered as "reversion". Those patients who have ASCUS, + HPV, LGSIL, or HGSIL on Pap smear at 11 to 15 months past their original Pap smear will be considered "persistent". Historical control subjects will also be grouped into "reversion" and "persistent" using the same criteria.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 26 years of age
* Women able to consent for themselves
* Referring Pap smear was ASCUS, + HPV or LGSIL
* Women who decide they wish to get the Gardasil vaccination series

Exclusion Criteria:

* Women who have had previous cryotherapy of the cervix, LEEP or cervical conization
* Women who had their first Gardasil injection prior to their referring Pap smear
* Women under the age of 18
* Women unable to consent for themselves
* Women who are pregnant currently trying to conceive
* Women in an immunocompromised state (diabetes, HIV, on chronic immunosuppressants or steroids, etc)
* Women who do not want the Gardasil vaccination series

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing colpo for initial low grade Pap abnormality who have elected to under Gardasil vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09-01 (Estimated); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean A. Seehusen, MD, MPH, Principal Investigator — Eisenhower Army Medical Center
Locations (1):
- Eisenhower Army Medical Center, Fort Gordon, Georgia, United States